CLINICAL TRIAL: NCT04305678
Title: Mepolizumab for the Treatment of Eosinophilic Fasciitis; An Open-Label, Single-Arm, Exploration Study
Brief Title: Mepolizumab for Eosinophilic Fasciitis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding lost from Sponsor.
Sponsor: Mayo Clinic (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Jason Sluzevich MD, Assistant Professor of Dermatology, College of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-011851
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Eosinophilic Fasciitis
Keywords: Mepolizumab
MeSH Terms: conditions — Eosinophilic Fasciitis | interventions — mepolizumab

STUDY DESIGN:
Intervention Model Description: Mepolizumab for the treatment of eosinophilic faciitis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Patients with a biopsy proven diagnosis of eosinophilic fasciitis
  Interventions: Drug: Mepolizumab

INTERVENTIONS:
Drug: Mepolizumab — Mepolizumab (Nucala) 400 mg SC every 4 weeks x 24 weeks
  Other Names: Nucala

SUMMARY:
This is a proof of concept pilot study to investigate the efficacy of mepolizumab in the treatment of eosinophilic fasciitis.

DETAILED DESCRIPTION:
This is an exploratory study designed to generate preliminary data in evaluating the efficacy of mepolizumab (Nucala) in the treatment of EF using mean change in the Rodnan Skin score (mRSS) before and after treatment. The study is powered at 90% to detect a 4 point change in the mRSS at a 5% significant level with a minimum target accrual of 6 patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years or older.
* History and physical examination consistent with EF
* Full thickness skin biopsy characteristic of eosinophilic fascitis and/or MRI radiographic findings characteristic of EF
* Documented peripheral eosinophilia (≥500 microliter)
* Patients who are willing and capable of cooperating to the extent and degree required by the protocol; and
* Patients who read and sign an approved informed consent for this study

Exclusion Criteria:

* Eosinophilic fascitis disease duration > 5 years
* Known history of adverse reaction to mepolizumab (Nucala)
* Pregnant females
* Females actively trying to conceive
* Vulnerable study population
* Asthma requiring inhaled cortiosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Modified Rodnan Skin Score (mRSS) | 24 weeks
  Mean change before and after treatment. The mRSS is a standardized scored assessment of tissue sclerosis as assessed by palpitation.

SECONDARY OUTCOMES:
Localized Scleroderma Skin Severity Index (mLoSSI) score | 24 weeks
  Mean change before and after treatment. mLoSSI score quantifies disease activity.
Localized Scleroderma Damage Index (LoSDI) score. | 24 weeks
  Mean change before and after treatment. LoSDI score quantifies disease damage.
Localized Scleroderma Cutaneous Assessment Tool (LoSCAT) | 24 weeks
  Mean change before and after treatment. LoSCAT is a composite score of disease activity (mLoSSI) and disease damage (LoSDI).
Physician's Global Assessment of Disease Activity (PhysGA-A) | 24 weeks
  Mean change before and after treatment. PhysGA-A is a 100-mm analog scale anchored by "inactive" at 0 and "markedly active" at 100.
Physician's Global Assessment of Disease Damage (PhysGA-D) | 24 weeks.
  Mean change before and after treatment. PhysGA-D is a 100-mm analog scale anchored by "no damage" at 0 and "markedly damaged" at 100.
Dermatology Quality of Life Index (DLQI) | 24 weeks.
  Mean change before and after treatment. DLQI is a skin-specific health questionnaire with higher scores reflecting decreased quality of life
Patient Global Assessment of Disease Severity (PtGA-S) | 24 weeks.
  Mean change before and after treatment.PhysGA-A is a 100-mm analog scale anchored by "not severe" at 0 and "very severe" at 100.

CONTACTS AND LOCATIONS:
Overall Officials: Jason C Sluzevich, M.D., Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials